CLINICAL TRIAL: NCT00990730
Title: Atherosclerosis in Rheumatoid Arthritis: Role of Inflammation, Lipoproteins, and Endothelial Dysfunction
Brief Title: Atherosclerosis in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Priscilla Hsue, Principle Investigator, University of California, San Francisco
Other Study IDs: H11397-34652-01; F32HL097461-01 (NIH); SFGH GCRC 6128
Record Dates: First submitted 2009-10-02; First posted 2009-10-07 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis; Endothelial Dysfunction
Keywords: rheumatoid arthritis; endothelial dysfunction; lipoproteins; inflammation; oxidative stress; arterial stiffness
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rheumatoid arthritis subjects: 60 subjects with rheumatoid arthritis, defined by American College of Rheumatology Criteria, enrolled in the UCSF RA cohort
- healthy controls: 20 matched controls without rheumatoid arthritis

SUMMARY:
The purpose of this study is to investigate the link between rheumatoid arthritis and cardiovascular disease by studying inflammation, joint disease, cholesterol abnormalities, and endothelial function.

DETAILED DESCRIPTION:
In the general population, individuals with elevated inflammatory markers (e.g. C-reactive protein, CRP) have increased cardiovascular disease. Patients with RA have chronic elevations in CRP and other inflammatory markers that are usually higher than the levels associated with increased cardiovascular risk in the general population. Indeed, RA patients have accelerated disease of their blood vessels, and increased cardiovascular death not explained by traditional cardiac risk factors but associated with chronic inflammation. However, the mechanisms by which inflammation leads to cardiovascular disease are not well characterized in RA. Moreover, current treatment strategies of RA largely target joint symptoms rather than inflammation, potentially leaving patients at increased risk for cardiovascular disease. Studies of markers that increase the risk of heart disease in the full spectrum of RA are missing. We hypothesize that inflammatory markers will be more strongly associated with abnormalities in blood vessels in RA patients than any clinical measure of disease activity. This hypothesis will be tested with a cross-sectional study of patients in the UCSF RA cohort. Aim 1 will characterize abnormal blood vessel changes across the spectrum of RA disease activity, specifically measuring ultrasound of the upper arm artery, markers of oxidative stress, and abnormalities in cholesterol proteins. Aim 2 will identify factors associated with these changes across the spectrum of RA disease activity, specifically focusing on the association between inflammatory markers, cholesterol, and blood vessel abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA by ACR criteria
* Age 18-80
* Enrolled in UCSF RA cohort already

Exclusion Criteria:

* Diabetes (on meds or in medical history)
* Pregnant or Lactating
* Renal failure (Creatinine > 2mg/dL or on dialysis)
* History of MI or CAD
* History of ischemic CVA
* Symptomatic PVD
* Current uncontrolled hypertension (blood pressure > 160/100mmHg)
* Daily prednisone > 10mg daily
* Current smoker
* New BP med within 3 months
* New statin within 3 months
* Change in RA meds: new or increase in prednisone within 1 month, new TNF inhibitor within 2 months, titration of methotrexate, leflunomide or sulfasalazine within 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: RA subjects are from the UCSF RA cohort based at San Francisco General Hospital and UCSF Medical Center. Controls will be selected from primary care clinics from these hospitals
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
flow mediated vasodilation of the brachial artery, measured by ultrasound | 1 day

SECONDARY OUTCOMES:
pulse wave velocity/arterial stiffness | day 1
lipid metabolism | day 1
pulse ampitude | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Y Hsue, MD, Principal Investigator — University of California, San Francisco; Peter Ganz, MD, Study Director — University of California, San Francisco
Locations (1):
- UCSF San Francisco General Hospital Vascular Research Center, San Francisco, California, United States